CLINICAL TRIAL: NCT00438750
Title: Prospective Randomized Comparison of Occupational Therapy vs Home Exercises After Volar Plate Fixation of a Fracture of the Distal Radius
Brief Title: Comparison of Occupational Therapy and Home Exercises for Adults With Operatively Treated Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator; Director of Research, Hand Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-001157
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Distal Radius Fractures
Keywords: distal radius fracture; rehabilitation; volar plate fixation; DASH questionnaire
MeSH Terms: conditions — Wrist Fractures | interventions — Occupational Therapy

ARMS (2):
- Independent Home Exercises (Experimental): Subjects who learn their therapy exercises from the surgeon and practice them independently at home.
  Interventions: Other: Independent Excercises
- Formal Therapy (Experimental): Subjects who follow the conventional protocol of seeing a therapist to learn and guide them in their exercises.
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Other: Independent Excercises — Subjects provided with wrist splint and instructions for independent exercises to perform at home on their own. Subjects were advised to perform exercises as often as possible, but at least three to four times a day for a minimum of thirty minutes. There was no formal strengthening program.
  Arms: Independent Home Exercises
Other: Occupational Therapy — Subjects were prescribed formal occupational therapy with supervised exercises to regain digit, wrist, and forearm motion and to strengthen the hand. The content, frequency, and duration of the rehabilitation program were at the discretion of the treating hand therapist.
  Arms: Formal Therapy

SUMMARY:
The purpose of this study is to compare to ways of rehabilitating after surgery for distal radius fractures treated operatively with a volar plate.

DETAILED DESCRIPTION:
Operative treatment of distal radius fractures has become commonplace over the last three decades as our understanding of the relationship between the alignment of the distal radius and the function of the wrist and forearm has improved. Over the last 15 years there has been a trend towards more invasive, internal plate fixation of fractures of the distal radius. One argument in favor of internal fixation for these fractures is that it would be beneficial to allow early movement of the wrist articulation in an attempt to maximize final outcome. There is a difference in opinion among physicians on the importance of supervision of exercises in the recovery process. Some physicians advocate formal occupational therapy while other physicians believe that appropriate instructions for home exercises are just as good. A common belief is that the motivation of the patient plays an important part in recovery. In addition, Psychological and personality factors, such as pain anxiety, catastrophizing, and depression are strongly related to upper extremity specific health status and may also influence recovery. The goal of this study is to determine which protocol for exercises leads to better outcome in patients treated for distal radius with a volar plate. As a secondary goal and to generate hypotheses for later studies we would like to evaluate the influence of psychosocial factors on both objective (motion, grip strength) and subjective (DASH questionnaire) measures of functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater.
* Isolated distal radial fracture.
* Fracture treated with volar plates, stable fixation.
* Initial treatment within 4 weeks of trauma.

Exclusion Criteria:

* Complex fractures that require additional or different material than volar plates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Independent Exercise Cohort: Subjects who learn their therapy exercises from the surgeon and practice them independently at home.
- Occupational Therapy Cohort: Subjects who follow the conventional protocol of seeing a therapist to learn and guide them in their exercises.
Period: Overall Study
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Started | 48 | 46
Completed | 39 | 37
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort | Total
Number analyzed (Participants) | 48 | 46 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 37 | 81
  >=65 years | 4 | 9 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (15) | 51 (15) | 50 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 48 | 46 | 94

OUTCOME MEASURES:

1. Primary Outcome: Range of Motion in Degrees of the Wrists
Description: Mean arc of wrist flexion and extension six months after surgery.
  Normal/expected range of motion for arc of wrist flexion and extension is approximately 160 degrees.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Number analyzed (Participants) | 39 | 37
Degrees | 129 (22.6) | 118 (17.7)

2. Secondary Outcome: Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire
Description: The DASH questionnaire measures arm-specific perceived disability. It contains 30 items and is scaled between zero and 100 with higher scores indicating worse upper-extremity function.
  Mean and standard deviations are identical for both arms.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Number analyzed (Participants) | 39 | 37
units on a scale | 7.8 (7.8) | 6.7 (6.7)

3. Secondary Outcome: 10-point Ordinal Pain Scale
Description: A ten point scale for pain at rest, with 0 as no pain and 10 as worst pain ever.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Number analyzed (Participants) | 39 | 37
units on a scale | 0.8 (1.4) | 1.0 (1.8)

4. Secondary Outcome: Pinch Strength
Description: Pinch strength measured with the B&L pinch gauge.
  B&L Engineering is the official name of the company (nowhere is there an expansion of this acronym).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Number analyzed (Participants) | 39 | 37
Pounds (lbs) | 15 (4.3) | 17 (8.6)

5. Secondary Outcome: Gartland and Werley Score
Description: An objective evaluation of wrist function with 0 to 2 as excellent, 3-8 as good, 9-20 as fair, and 21 and above as poor range of motion.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Number analyzed (Participants) | 39 | 37
units on a scale | 0.9 (1.2) | 1.1 (1.3)

6. Secondary Outcome: Mayo Wrist Score
Description: A composite score based on pain intensity, range of motion, grip strength, and functional status. The scale is as follows: below 60 is poor, 60-80 is satisfactory, 80-90 is good, and 90-100 is excellent.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Number analyzed (Participants) | 39 | 37
units on a scale | 83.4 (12.7) | 79.0 (9.9)

7. Secondary Outcome: Grip Strength
Description: Measured with use of a grip meter as the average of three attempts.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Number analyzed (Participants) | 39 | 37
Pounds (lbs) | 57 (18.5) | 51 (17.9)

ADVERSE EVENTS:
Arm/Group | Independent Exercise Cohort | Occupational Therapy Cohort
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/46
Other Adverse Events (participants affected / at risk) | 0/48 | 2/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Independent Exercise Cohort (N=48) | Occupational Therapy Cohort (N=46)
Extensor pollicis longus tendon rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Subject declined tendon transfer
Loosening and prominence of a distal (periarticular) screw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Subject underwent implant removal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No